CLINICAL TRIAL: NCT00243776
Title: Molecular and Cellular Characterization of Cardiac Tissue in Postnatal Development
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Davis, Associate Professor, Emory University
Other Study IDs: IRB00005500; R01HL077485 (NIH); 35328 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Disease; Tetralogy of Fallot
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue obtained from surgical waste tissue
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Cardiac Tissue: Cardiac tissue and cells will be obtained from participants undergoing cardiac surgical repair

SUMMARY:
The study team will use small pieces of human hearts which are removed as part of a required surgical procedure to study different objectives. One of the objective is how calcium ions pass through the membrane of heart cells in order to tell the heart cell how much force to contract with when the heart beats. Investigators will also study the proteins and RNA of these pieces to determine how the newborn heart cells control their force of contraction differently from adult heart cells. Investigators hypothesize that infant hearts have different regulation of calcium entry than adult hearts. The study team also wants to study combinations of 3D cardiac spheres with multiple environmental cues that can improve functional and metabolic maturation of Human pluripotent stem cell-derived cardiomyocytes (hPSC-CMs) and generate a more clinically relevant cell model.

DETAILED DESCRIPTION:
Extrapolating pharmacological and surgical therapies from adult (AD) studies to infant (INF) patients is problematic because the knowledge of cellular electrophysiology and molecular biology of human INF heart cells is limited. The investigators have studied developmental differences in rabbit ventricular cells and now extend these studies to atrial and ventricular cells isolated from AD, young adult (YAD) or INF patients.

The study aims are as follows:

1. Developmental differences in transient outward current of atrial cells. Investigators will extend their studies to isolated cells and tissue from YADs (age 14-20). In addition, several other accessory beta-subunits have been found in cardiac myocytes and may interact with Kv channels and regulate the function of these channels. The study team will determine relative amounts of these putative regulators of human atrial Ito to determine which correlate with developmental changes in Ito kinetics.
2. Developmental differences in amplitude and regulation of calcium current in atrial cells. Investigators hypothesize that INF atrial cells have tonic inhibition of adenylyl cyclase (and thus of ICa) mediated by inhibitory G proteins, possibly related to constitutive activity of the adenosine A1 receptor, and that, compared to AD or YAD cells, have greater sensitivity to inhibitors of phosphatases and phosphodiesterases, and that developmental changes in basal ICa amplitude and beta-sympathetic modulation correlate with inhibitory G protein levels, receptor numbers for M2 and A1 receptors, and constitutive inhibitory activity.
3. Modulation of atrial cell calcium transients by changes in AP waveform and developmental age. The study team will test the hypothesis that prolongation of the early repolarization phase of the after potential (AP) increases Ca2+ entry and that YAD cells have faster removal of Ca2+ from cytoplasm than INF cells and will determine if the Na- Ca2+ exchange current (INCX) is greater in INF vs. AD or YAD cells.
4. Developmental differences in Ca current and transients and contractility in ventricular cells. Investigators propose that INF cells and tissue have lower basal ICa, lower potency for Isoproterenol stimulation, higher levels of Gialpha3 and A1 receptors, greater inhibitory potency for adenosine, and tonic inhibition of ICa. We also propose that the YAD cells have lower levels of NCX and lower INCX, higher levels of SERCA and faster removal of Ca2+ from the cytoplasm. Previous animal studies have indicated various developmental changes in cardiac cells. We will specifically study human postnatal developmental changes in Ito, regulation of ICa and intracellular Ca2+ transients.
5. Structural, Functional and Metabolic Maturation of hPSC-CMs. Investigators propose that combinations of 3D cardiac spheres with multiple environmental cues to improve mitochondrial fatty acid oxidation (FAO or beta-oxidation) pathway will promote functional and metabolic maturation of hPSC-CMs and generate a more clinically relevant model. using tissue engineering combined with pharmacological agents to regulate signals that are involved in FAO metabolism and appropriate growth factor and hormonal signaling that mimic the microenvironment for the maturation of CMs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiopulmonary bypass surgery
* Patients undergoing surgery for repair of congenital heart disease such as ventricular septal defect or defective mitral or aortic valves.

Exclusion Criteria:

* Prior cardiac surgery
* History of atrial fibrillation or other atrial arrhythmias prior to operation
* History of heart failure

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing surgery for repair of congenital heart disease
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2005-04; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Calcium Current Measures | Duration of Study (Up to 13 Years)
  Calcium currents including transients and modulation of calcium handling by activation of different pathways in isolated cells from waste tissue obtained at the time of surgical repair for Congenital Heart Disease will be measured for the duration of the study.
Change in structural, functional and metabolic maturation of Human pluripotent stem cell derived Cardiomyocytes (hPSC-CMs) | Duration of Study (Up to 3 Years)
  Change in structural, functional and metabolic maturation of Human pluripotent stem cell derived Cardiomyocytes (hPSC-CMs) is achieved using combinations of 3D cardiac spheres with multiple environmental cues to improve mitochondrial fatty acid oxidation (FAO or beta-oxidation) pathway will promote functional and metabolic maturation of hPSC-CMs and generate a more clinically relevant model. The outcome will be measured whether the cells achieved maturation (structural, functional and metabolic maturation) or not after using combinations of 3D cardiac spheres with multiple environmental cues.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Davis, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wiegerinck RF, Cojoc A, Zeidenweber CM, Ding G, Shen M, Joyner RW, Fernandez JD, Kanter KR, Kirshbom PM, Kogon BE, Wagner MB. Force frequency relationship of the human ventricle increases during early postnatal development. Pediatr Res. 2009 Apr;65(4):414-9. doi: 10.1203/PDR.0b013e318199093c. PMID 19127223